CLINICAL TRIAL: NCT03824652
Title: WALNUTS for POWER: Polyphenols, Omega-3 Fatty Acids, Weight Loss, and EneRgy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Freedland (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor-Investigator, Stephen Freedland, Professor, Surgery, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018-23-Freedland-POWR
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate adenocarcinoma; diet; walnuts; radical prostatectomy; omega-3 fatty acids; polyphenols
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Diet + Walnuts (Experimental): Usual diet with the addition of two ounces of walnuts daily, phone counseling with dietitian, for 4-10 weeks
  Interventions: Other: walnuts; Other: usual diet; Other: phone counseling with dietitian
- Usual Diet (Active Comparator): Usual diet for 4-10 weeks
  Interventions: Other: usual diet

INTERVENTIONS:
Other: walnuts — 2 ounces of walnuts daily for 4-10 weeks
  Arms: Usual Diet + Walnuts
Other: usual diet — Subject continues usual diet
Other: phone counseling with dietitian — Weekly calls with dietitian
  Arms: Usual Diet + Walnuts

SUMMARY:
This is a randomized control trial testing the effect of walnut supplementation on prostate cancer progression in 50 men with biopsy confirmed prostate cancer and planning to undergo RP. Patients consented to the study will be randomly assigned to either continue their usual diets (control arm) or to the walnut arm for 4-10 weeks depending on the window between their consent date and the date for RP.

DETAILED DESCRIPTION:
The overall objective of this study is to test the effect of walnuts added to a usual diet on prostate cancer progression as measured by Ki67 expression in the prostate tissues. Subjects will be randomized 1:1 to usual diet or usual diet with the addition of 2 ounces of walnuts daily. The baseline visit will occur in conjunction with a standard of care visit post-biopsy, the intervention period will range from 4-10 weeks dependent upon the scheduled date of the standard of care radical prostatectomy (RP), and the final visit will occur in conjunction with a standard of care visit prior to RP.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed prostate adenocarcinoma.
* Diagnostic biopsy cores with ≥10 cores with each core examined separately to determine exact tumor location.
* Biopsy grade group 2 or higher (Gleason ≥7).
* Planning to undergo RP.
* Willing to adhere to a usual diet with the possible addition of 2 oz of walnuts per day.
* Reads, writes, and understands English.
* Age 18 or older

Exclusion Criteria:

* Allergy to nuts.
* History of receiving hormone therapy or antiandrogen therapy.
* Use of 5-alpha reductase inhibitors in the past 6 months.
* Prior prostate radiotherapy (external beam or brachytherapy) or prior prostate cryotherapy.
* Currently enrolled in a modified diet/weight loss program and/or taking dietary supplements that contain omega-3s (e.g., fish oil).
* Other active malignancy, excluding basal cell carcinoma or squamous cell carcinoma
* Significant co-morbidities (e.g., cardiac, pulmonary, liver disease, alcohol/drug addiction, malabsorption syndromes), that in the opinion of the study physician make the patient ineligible.
* Individuals with psychological/mental conditions which can affect the consent process and/or their adherence to the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean difference in prostatic tissue Ki67 expression from baseline biopsy to RP | 10 weeks

SECONDARY OUTCOMES:
Mean difference in prostatic tissue oxidative stress from baseline biopsy to RP | 10 weeks
  Measured by prostate tissue 8-hydroxy-2-deoxyguanosine
Mean difference in prostatic tissue inflammation from baseline biopsy to RP | 10 weeks
  Measured by 8-hydroxy-2-deoxyguanosine and immune cell infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedland, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Durham VA Medical Center, Durham, North Carolina